CLINICAL TRIAL: NCT06842693
Title: Evaluating Chile's Proposed Non-nutritive Sweeteners Warning Label Regulation
Brief Title: Testing Non-nutritive Sweetener Labels in Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other); Bloomberg Philanthropies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-2896a; 24-2205 (Other Grant/Funding Number: Bloomberg Philanthropies)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Behavioral: Control
- Chilean non-nutritive sweetener label (Experimental)
  Interventions: Behavioral: Chilean non-nutritive sweetener label
- Colombian non-nutritive sweetener label (Experimental)
  Interventions: Behavioral: Colombian non-nutritive sweetener label

INTERVENTIONS:
Behavioral: Control — Products carry neutral control label when containing non-nutritive sweeteners. Additionally, to match the current Chilean legislation, products carry an octagonal label that states "high in sugar" when high in added sugars, and/or an octagonal label that states "high in calories" when high in calorie density.
  Arms: Control
Behavioral: Chilean non-nutritive sweetener label — Products carry rectangular label that states "contains non-nutritive sweeteners, not recommended for children" when containing non-nutritive sweeteners. Additionally, to match the current Chilean legislation, products carry an octagonal label that states "high in sugar" when high in added sugars, and/or an octagonal label that states "high in calories" when high in calorie density.
  Arms: Chilean non-nutritive sweetener label
Behavioral: Colombian non-nutritive sweetener label — Products carry octagonal label that states "contains non-nutritive sweeteners " when containing non-nutritive sweeteners. Additionally, to match the current Chilean legislation, products carry an octagonal label that states "high in sugar" when high in added sugars, and/or an octagonal label that states "high in calories" when high in calorie density.
  Arms: Colombian non-nutritive sweetener label

SUMMARY:
The goal of this experiment is to examine the effects of 2 types of non-nutritive sweetener (NNS) warning labels among a sample of Chilean parents. The main questions this experiment aims to answer are:

Do non-nutritive sweetener warning labels improve consumers' ability to identify when a product contains non-nutritive sweeteners?

Do non-nutritive sweetener warning labels impact on consumers' selection of non-nutritive sweetener-sweetened, unsweetened, and/or sugar-sweetened products for their children?

Participants will be randomly assigned to 1 of 3 types of labels and view their assigned label on 3 sets of products. Each set will display 4 similar products: one unsweetened, one sweetened with sugar, one sweetened with non-nutritive sweeteners, and one sweetened with both sugar and non-nutritive sweeteners. For each set, participants will identify which product(s) contain NNS and select the product that they would purchase for their child. Researchers will compare results across label types.

DETAILED DESCRIPTION:
Participants will complete an online randomized experiment programmed in Qualtrics. After providing informed consent, participants will be randomly assigned to view 1 of 3 types of labels: a neutral control label, a rectangular label stating "contains non-nutritive sweeteners, not recommended for children" (i.e., Chilean NNS label), or an octagonal label stating "contains non-nutritive sweeteners" (i.e., Colombian NNS label).

Participants will view their assigned label on 4 similar products (one unsweetened, one sweetened with sugar, one sweetened with non-nutritive sweeteners, and one sweetened with both sugar and non-nutritive sweeteners) displayed in random order and complete a task where they identify which product(s) contain non-nutritive sweeteners and select one of the products to purchase for their child. During this task, in all arms, products will also display Chile's current nutrient warning labels when applicable. This task will be repeated 3 times, each time with a different product category (i.e., fruit drinks, yogurts, breakfast cereals), with categories displayed in random order.

After the selection/identification tasks, participants will view their assigned labels on 2 products containing non-nutritive sweeteners (i.e., flavored milk and cereal bar). For each product, participants will rate the perceived message effectiveness of the label and perceived product healthfulness. Lastly, after all product exposures, participants will rate their intentions to limit their child's non-nutritive sweetener consumption.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Parent or guardian of child between 2-14 years old who has never been diagnosed with diabetes, high blood sugar, pre-diabetes or insulin resistance
* Residing in Chile

Exclusion Criteria:

* Less than 18 years old
* Not parent or guardian of child between 2-14 years old who has never been diagnosed with diabetes, high blood sugar, pre-diabetes or insulin resistance
* Not residing in Chile

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3916 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Correct identification of non-nutritive sweetener containing products | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Correct identification of products that contain non-nutritive sweeteners will be measured by survey. Response will be coded in a dichotomous 0-1 range, where 1 indicates that the participant correctly identified the products that contained non-nutritive sweeteners and 0 indicates that the participant did not correctly identify the products that contained non-nutritive sweeteners.
Selection of non-nutritive sweetener-sweetened product for purchase | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Selection of sugar-sweetened product for purchase will be measured by survey. Response will be coded in a dichotomous 0-1 range, where 1 indicates that the participant chose one of the non-nutritive sweetener-sweetened products and 0 indicates that the participants selected one of the other two products.
Selection of unsweetened product for purchase | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Selection of unsweetened product for purchase will be measured by survey. Response will be coded in a dichotomous 0-1 range, where 1 indicates that the participant chose the unsweetened product and 0 indicates that the participants selected one of the other three products.
Selection of sugar-sweetened product for purchase | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Selection of sugar-sweetened product for purchase will be measured by survey. Response will be coded in a dichotomous 0-1 range, where 1 indicates that the participant chose one of the sugar-sweetened products and 0 indicates that the participants selected one of the other two products.

SECONDARY OUTCOMES:
Perceived message effectiveness, mean score | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Perceived message effectiveness will be measured by survey through a three-item scale. Items will inquire about how much participants perceive the label to (1) discourage them from wanting to buy products with non-nutritive sweeteners for their child, (2) makes them concerned about the health effects of their child consuming products with non-nutritive sweeteners, and (3) makes buying products with non-nutritive sweeteners for their child seem unpleasant to them. Response options will be on a 5-point scale between "not at all" (coded as 1) and "very much" (coded as 5), with higher scores representing a higher perceived message effectiveness. Each participant's responses to each item will be combined to obtain their final score on the outcome.
Perceived product healthfulness, mean score | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  How good or bad for participants' children it would be to consume the product every day will be measured by survey. Response options will be on a 5-point scale between "very bad" (coded as 1) and "very good" (coded as 5), with higher scores representing a higher perceived product healthfulness.
Relative product healthfulness, mean score | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  How healthy participants perceive the non-nutritive sweetener-containing product to be compared to the version of the product that contains added sugars will be measured by survey. Response options will be on a 5-point scale between "much less healthy" (coded as 1) and "much healthier" (coded as 5), with higher scores representing a higher comparative product healthfulness.
Intentions to limit non-nutritive sweetener consumption, mean score | After exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  How much participants intend to limit their child's consumption of non-nutritive sweeteners in the next week will be measured by survey. Response options will be on a 5-point scale between "not at all" (coded as 1) and "very much" (coded as 5), with higher scores representing a higher intention to limit consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Smith Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill's Gillings School of Global Public Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared prior to data collection. After data collection and analysis, a de-identified version of individual participant data and the analytic code will be shared through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol and statistical analysis plan will be available by March 2025 (prior to data collection). A de-identified version of the data collected and analytic code used will become available after data collection and analysis and will remain available indefinitely.
Access Criteria: Open access
URL: https://osf.io/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT06842693/Prot_SAP_000.pdf